CLINICAL TRIAL: NCT05096663
Title: A Phase II/III Study of N-803 (ALT-803) Plus Pembrolizumab Versus Standard of Care in Participants With Stage IV or Recurrent Non-Small Cell Lung Cancer Previously Treated With Anti-PD-1 or Anti-PD-L1 Therapy (Lung-MAP Non-Match Sub-Study)
Brief Title: Testing the Use of Combination Immunotherapy Treatment (N-803 [ALT-803] Plus Pembrolizumab) Against the Usual Treatment for Advanced Non-small Cell Lung Cancer (A Lung-MAP Treatment Trial)
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1800D; NCI-2021-09852 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1800D (Other: SWOG); S1800D (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Advanced Lung Non-Small Cell Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Vitamin B 12; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Docetaxel; Folic Acid; Leucovorin; Gemcitabine; ALT-803; pembrolizumab; Pemetrexed; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (standard of care) (Active Comparator): Patients receive standard of care consisting of docetaxel IV over 30-60 minutes on day 1; gemcitabine IV over 30 minutes on days 1 and 8; pemetrexed IV over 10 minutes on day 1; or ramucirumab IV over 30-60 minutes and docetaxel IV over 30-60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: Cobalamin; Drug: Dexamethasone; Drug: Docetaxel; Dietary Supplement: Folic Acid; Drug: Gemcitabine; Drug: Pemetrexed; Biological: Ramucirumab
- Arm B (pembrolizumab, nogapendekin alfa) (Experimental): Patients receive pembrolizumab IV over 30 minutes and nogapendekin alfa SC on day 1. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients then receive nogapendekin alfa SC on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Nogapendekin Alfa; Biological: Pembrolizumab

INTERVENTIONS:
Dietary Supplement: Cobalamin — Given intramuscularly
  Other Names: B12 Vitamin; Cobalamin (1+); VIT B12; Vitamin B-12; Vitamin B12; Vitamin-B12
  Arms: Arm A (standard of care)
Drug: Dexamethasone — Given orally (PO)
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
  Arms: Arm A (standard of care)
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Arm A (standard of care)
Dietary Supplement: Folic Acid — Given PO
  Other Names: 2-[4-[(2-amino-4-oxo-1H-pteridin-6-yl)methylamino]benzoyl]aminopentanedioic acid; FA; Folacin; Pteroylmonoglutamic Acid; Vitamin B9; Vitamin Bc
  Arms: Arm A (standard of care)
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
  Arms: Arm A (standard of care)
Drug: Nogapendekin Alfa — Given SC
  Other Names: ALT 803; ALT-803; ALT803; Fusion Protein Consisting of IL-15N72D and IL-15RaSu/FC; IL-15N72D/IL-15Ra-Fc; IL-15N72D:IL-15RaSu/Fc Fusion Complex; N 803; N-803; N803; Superagonist Interleukin-15:Interleukin-15 Receptor AlphaSu/Fc Fusion Complex Alt-803
  Arms: Arm B (pembrolizumab, nogapendekin alfa)
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
  Arms: Arm B (pembrolizumab, nogapendekin alfa)
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate; Pemfexy
  Arms: Arm A (standard of care)
Biological: Ramucirumab — Given IV
  Other Names: Anti-VEGFR-2 Fully Human Monoclonal Antibody IMC-1121B; Cyramza; IMC-1121B; LY3009806; Monoclonal Antibody HGS-ETR2
  Arms: Arm A (standard of care)

SUMMARY:
This phase II/III Lung-MAP trial studies how well immunotherapy treatment with N-803 (ALT-803) and pembrolizumab working in treating patients with non-small cell lung cancer that has spread to other places in the body (advanced). Natural killer cells, part of our immune system, are always on alert and ready to defend our bodies from many kinds of infection or rogue cells, such as those that cause cancer. N-803 (ALT-803) may activate natural killer cells so that they can stimulate an immune response to help fight cancer. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving N-803 (ALT-803) and pembrolizumab may help shrink and stabilize lung cancer or prevent it from returning.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare overall survival (OS) between participants randomized to nogapendekin alfa (N-803 [ALT-803]) + pembrolizumab versus standard of care therapy. (Primary Resistance Cohort) II. To compare overall survival (OS) between participants randomized to N-803 (ALT-803) + pembrolizumab versus standard of care therapy. (Acquired Resistance Cohort)

SECONDARY OBJECTIVES:

I. To compare investigator assessed progression-free survival (IA-PFS) with confirmation of progression by immune response criteria between the treatment arms.

II. To compare investigator assessed progression-free survival (IA-PFS) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 between the treatment arms.

III. To compare the response rates between the arms. IV. To evaluate duration of response (DoR) among responders. V. To evaluate the frequency and severity of toxicities within each treatment arm.

TRANSLATIONAL MEDICINE OBJECTIVE:

I. To establish a blood repository to pursue future studies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive standard of care consisting of docetaxel intravenously (IV) over 30-60 minutes on day 1; gemcitabine IV over 30 minutes on days 1 and 8; pemetrexed IV over 10 minutes on day 1; or ramucirumab IV over 30-60 minutes and docetaxel IV over 30-60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive pembrolizumab IV over 30 minutes and nogapendekin alfa subcutaneously (SC) on day 1. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients then receive nogapendekin alfa SC on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been assigned to S1800D by the Southwest Oncology Group (SWOG) Statistics and Data Management Center (SDMC). Assignment to S1800D is determined by the LUNGMAP or S1400 protocol
* Participants must have measurable or non-measurable disease documented by computed tomography (CT) or magnetic resonance imaging (MRI). Measurable disease must be assessed within 28 days prior to randomization. Non-measurable disease must be assessed within 42 days prior to randomization. The CT from a combined positron emission tomography (PET)/CT may be used only if it is of diagnostic quality. All known sites of disease must be assessed and documented on the Baseline Tumor Assessment Form (RECIST 1.1)
* Participants must have a CT or MRI scan of the brain to evaluate for central nervous system (CNS) disease within 42 days prior to sub-study randomization
* Participants with spinal cord compression or brain metastases must have received local treatment to these metastases and remained clinically controlled and asymptomatic for at least 7 days following stereotactic radiation and/or 14 days following whole brain radiation, and prior to sub-study randomization
* Participants with spinal cord compression or brain metastases must not have residual neurological dysfunction, unless no further recovery is expected, and the participant has been stable on weaning doses of corticosteroids (=< 10 mg daily prednisone or equivalent) prior to sub-study randomization
* Participants must have progressed (in the opinion of the treating investigator) following the most recent line of therapy for non-small cell lung cancer (NSCLC)
* Participants with a known sensitizing mutation for which an FDA-approved targeted therapy for NSCLC exists (e.g. EGFR, ALK gene fusions, ROS1, BRAF, RET, NTRK, and MET sensitizing mutations), must have previously received at least one of the approved therapy(s)
* Participants must have received exactly one line of anti-PD-1 or anti-PD-L1 therapy for advanced disease (stage IV or recurrent, or stage III in certain circumstances outlined below) given alone or in combination with platinum-based chemotherapy. Participants must have experienced disease progression during or after this regimen

  * Continuing the same agent(s) after progression counts as a single line of therapy. However, a change or addition in agent(s) after progression (e.g. the addition of chemotherapy to anti-PD-1 monotherapy after progression) counts as a subsequent line of therapy and would exclude the participant
  * For participants who received consolidation anti-PD-1 or anti-PD-L1 therapy following concurrent chemoradiation for Stage III disease as their only line of anti-PD-1 or anti-PD-L1 therapy:

    * If they experienced disease progression less than (<) 365 days from the first date of anti-PD-1 or anti-PD-L1 therapy, this counts as the single line of anti-PD-1 or anti-PD-L1 therapy for advanced disease
    * If they experienced disease progression more than or equal to (>=) 365 days from the first date of anti-PD-1 or anti-PD-L1 therapy, this is not considered a line of anti-PD-1 or anti-PD-L1 therapy for advanced disease
* Participants must have recovered (=< grade 1) from any side effects of prior therapy, except for alopecia
* Participants must be able to safely receive at least one of the investigator's choice of standard of care regimens, per the current FDA-approved package insert

  * Note: Pemetrexed is not FDA-approved for squamous cell NSCLC and must not be used to treat participants with squamous cell NSCLC
* Absolute neutrophil count (ANC) >= 1.5 x 10^3/uL (obtained within 28 days prior to sub-study randomization)
* Platelet count >= 100 x 10^3/uL(obtained within 28 days prior to sub-study randomization)
* Hemoglobin >= 9 g/dL (obtained within 28 days prior to sub-study randomization)
* Serum bilirubin =< institutional upper limit of normal (IULN) (within 28 days prior to sub-study randomization). For participants with liver metastases, bilirubin must be =< 5 x IULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2 x IULN (within 28 days prior to sub-study randomization). For participants with liver metastases, ALT and AST must be =< 5 x IULN
* Serum creatinine =< the IULN or calculated creatinine clearance >= 50 mL/min using Cockcroft-Gault formula. This specimen must have been drawn and processed within 28 days prior to sub-study randomization
* Participants' most recent Zubrod performance status must be 0-1 and be documented within 28 days prior to sub-study randomization
* Participants must have history and physical exam must be obtained within 28 days prior to sub-study randomization
* Participants with known human immunodeficiency virus (HIV) infection must be receiving anti-retroviral therapy and have an undetectable viral load at their most recent viral load test within 6 months prior to sub-study randomization
* Participants must also be offered participation in banking and in the correlative studies for collection and future use of specimens
* Note: As a part of the OPEN registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

  * Participants must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines

Exclusion Criteria:

* Participants must not have leptomeningeal disease that requires CNS-specific treatment prior to registration and must not be planning to receive the CNS-specific treatment through the first cycle of the protocol therapy
* Participants must not have experienced the following:

  * Any grade 3 or worse immune-related adverse event (irAE). Exception: asymptomatic nonbullous/nonexfoliative rash
  * Any unresolved grade 2 irAE
  * Any toxicity that led to permanent discontinuation of prior anti-PD-1/PD-L1 immunotherapy
  * Exception to the above: Toxicities of any grade that requires replacement therapy and has stabilized on therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) are allowed
* Participants must not have any history of organ transplant that requires use of immunosuppressives
* Participants must not have history of (non-infectious) pneumonitis that required steroids or current pneumonitis/interstitial lung disease
* Participants must not have any known allergy or reaction to any component of the investigational formulations. If there is a known allergy or reaction to standard of care formulations, participants must be able to safely receive at least one of the standard of care options
* Participants must not have any grade III/IV cardiac disease as defined by the New York Heart Association Criteria (i.e., participants with cardiac disease resulting in marked limitation of physical activity or resulting in inability to carry on any physical activity without discomfort), unstable angina pectoris, and myocardial infarction within 6 months prior to sub-study randomization, or serious uncontrolled cardiac arrhythmia
* Participants must not have experienced any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to sub-study randomization
* Participants must not have an active or uncontrolled infection in the opinion of the treating investigator
* Participants must not have a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Participants must not have any of following:

  * Cirrhosis at a level of Child-Pugh B (or worse)
  * Cirrhosis (any degree) and a history of hepatic encephalopathy
  * Or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis
* Participants must not have received anti-CTLA4 therapy (e.g. ipilimumab, tremelimumab), or other immune-modulatory therapy (e.g. anti-TIM-3, anti-LAG-3, anti-GITR, IL-2, IL-15)
* Participants must not have received any prior systemic therapy (systemic chemotherapy, immunotherapy or investigational drug) within 21 days prior to sub-study randomization
* Participants must not have received any radiation therapy within 14 days prior to sub-study randomization
* Participants must not have received nitrosoureas or mitomycin-c within 42 days prior to sub-study randomization
* Participants must not have received systemic treatment with corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 7 days prior to sub-study randomization. Inhaled or topical steroids, and adrenal replacement doses =< 10 mg daily prednisone or equivalent are permitted in the absence of active autoimmune disease
* Participants must not have received a live attenuated vaccination within 28 days prior to sub-study randomization. All COVID-19 vaccines that have received Food and Drug Administration (FDA) approval or FDA emergency use authorization are acceptable
* Participants must not be planning to receive any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment while receiving treatment on this study
* Participants must not have had a major surgery within 14 days prior to sub-study randomization. Participant must have fully recovered from the effects of prior surgery in the opinion of the treating investigator
* Participants must not have an active autoimmune disease that has required systemic treatment within two years prior to sub-study randomization (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
* Participants must not have any history of primary immunodeficiency
* Participants must not be pregnant or nursing. Women/men of reproductive potential must have agreed to use an effective contraceptive method during the study and 4 months after completion of study treatment. A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. However, if at any point a previously celibate participant chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures during the study and 4 months after study completion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to 2 years
  Will be compared between the arms using the combination weighted/unweighted log-rank test statistic (as utilized in S1800A) with statistical significance at the 1-sided 10% level.

SECONDARY OUTCOMES:
Investigator-assessed progression-free survival (IA-PFS) | From date of sub-study randomization to date of first documentation of potential immune-response confirmed progression, or death due to any cause, assessed up to 2 years
  Will be compared between the arms using the combination weighted/unweighted log-rank test statistic (as utilized in S1800A) with statistical significance at the 1-sided 10% level.
Duration of response (DoR) | From date of first documentation of response (complete response or partial response) to date of first documentation of progression assessed by local review or symptomatic deterioration, or death due to any cause, assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John M Wrangle, Principal Investigator — SWOG Cancer Research Network
Locations (350):
- United States (350):
  - Veterans Administration Medical Center - Birmingham, Birmingham, Alabama
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe South Coastal Health Campus, Frankford, Delaware
  - Bayhealth Hospital Sussex Campus, Milford, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Mercyhealth Javon Bea Hospital - Rockton, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - HaysMed University of Kansas Health System, Hays, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Kaiser Permanente-Woodlawn Medical Center, Baltimore, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente - Kensington Medical Center, Kensington, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Ascension Providence Hospitals - Novi, Novi, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Cancer Institute at Saint Francis Hospital, East Hills, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - University of Rochester, Rochester, New York
  - Good Samaritan Hospital Medical Center, West Islip, New York
  - Randolph Hospital, Asheboro, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - AdventHealth Infusion Center Weaverville, Weaverville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - UPMC Hillman Cancer Center at Butler Health System, Butler, Pennsylvania
  - UPMC Camp Hill, Camp Hill, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Chambersburg, Pennsylvania
  - UPMC Hillman Cancer Center - Passavant - Cranberry, Cranberry Township, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Oncology Hematology Associates, Greenville, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - UPMC Hillman Cancer Center - Part of Frick Hospital, Mount Pleasant, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - UPMC Cancer Center-Natrona Heights, Natrona Heights, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC-Mercy Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center-Uniontown, Uniontown, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - UPMC West Mifflin-Cancer Center Jefferson, West Mifflin, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Kaiser Permanente-Burke Medical Center, Burke, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin